CLINICAL TRIAL: NCT01441752
Title: State Administration of Traditional Chinese Medicine of Shanghai
Brief Title: Efficacy Study of Integrated TCM Combined With Chemotherapy in Postoperative NSCLC Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: xuling (Other)
Responsible Party: Sponsor-Investigator, xuling, State Administration of Traditional Chinese Medicine of Shanghai, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC 001
Record Dates: First submitted 2011-07-14; First posted 2011-09-28 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + TCM group (Experimental): The chemotherapy for NSCLC patients is a combination of Vinorelbine, 25mg/m2, d1, 8 and DDP, 75mg/m2, d1 (NP) giving three-weekly for four cycles.
  Prescriptions formulated into granules origin from Professor Liu Jiaxiang in Longhua hospital. Package of granules is made into three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe . Each package contained 20g of water-soluble herbal granules that were manufactured at a Good Manufacture Practice standard facility (Tian Jiang Ltd, Jiangyin, China). Each package was labeled with a serial number. The prescription form comprised the stock list with both the name and serial number.
  Interventions: Drug: TCM
- Chemotherapy + placebo group (Placebo Comparator): The chemotherapy for NSCLC patients is a combination of Vinorelbine, 25mg/m2, d1, 8 and DDP, 75mg/m2, d1 (NP) giving three-weekly for four cycles.we compromise the raw materials for the placebo including 10% of Chinese medicine, food color and artificial flavors. The placebo and therapeutic packages were stored in different cabinets, and only the dispensing technician knew the contents of the packages.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TCM — three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe.
  Other Names: Prescriptions from Professor Liu Jiaxiang
  Arms: Chemotherapy + TCM group
Drug: placebo — three types with functions such as benefiting Qi recipe, benefiting Yin recipe and detoxication and resolving masses recipe，with the same color, smell ，taste weight and package
  Arms: Chemotherapy + placebo group

SUMMARY:
The investigators performed a multi-center, randomized, controlled, double-blind, prospective study on evaluating effect of chemotherapy combined with or without integrated TCM on quality of life (QOL) of postoperative Non-small Cell Lung Cancer (NSCLC) patients. The investigators plan to involve 600 cases for observation in 3 years (300 cases for each group), expecting that QOL of postoperative NSCLC patients can be improved by integrated TCM combined with chemotherapy compared to that by chemotherapy alone.

DETAILED DESCRIPTION:
At present the high rate of recurrence and metastasis of postoperative non-small cell lung cancer (NSCLC) patients is one of the leading causes resulting in failure of treating lung cancer. More than 35% of postoperative lung cancer patients with stage I died in 5 years due to recurrence or metastasis; the 5-year survival rates of stage II, IIIa, IIIb were 31%, 17.9% and 11.7% respectively. The survival rate was improved by 5% with adjuvant chemotherapy after resection, so regimen consist of platinum-based two chemical medicines are commended as the adjuvant chemotherapy for treating postoperative NSCLC patients, but the toxicity and side effects of chemotherapy can decrease quality of life (QOL) of patients. Literature and our preliminary studies have shown that traditional Chinese medicine (TCM) can prolong survival and improve QOL, but high-level evidences are needed.

The investigators perform a randomized, double-blind study in NSCLC patients after complete resection with stage I-III. Patients are randomized over observational group (TCM granules plus chemotherapy), and control group (TCM placebo plus chemotherapy). The investigators will observe 4 treatment periods, after that the observational group will be treated for another 4 months with integrated TCM combined with western medicine treatment (oral TCM medicines plus TCM intravenous injections), and there is no intervene measures in control group. Regular follow-up will be arranged. The primary efficacy assessments are: QOL (QLQ-C30 scales); Secondary efficacy assessments are: (1) 2-year disease-free survival rate; (2) disease-free survival; other efficacy assessments are: (1) TCM symptoms changes; (2) tumor markers (CEA, CA-125 and CYFRA21-1) and so on. Toxicity, side effects and security of the treatments will be assessed at the same time. The investigators expect that integrated TCM combined with Western medicine treatment has a better efficacy on improving QOL of patients, prolonging disease-free survival time than that of chemotherapy treatment. Therefore our study can provide evidences for optimizing and promoting integrated TCM combined with Western Medicine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of primary bronchial lung cancer, and pathologically or cytologically confirmed of NSCLC (squamouscarcinoma, adenocarcinoma, adenosquamous carcinoma and large cell carcinoma) patients;
2. Age > 18 years old;
3. TCM syndromes are Yin deficiency, Qi deficiency, deficiency of both Qi and Yin, deficiency of both Spleen and Kidney;
4. Physical status score (ECOG PS) ≤ 2 scores;
5. Stage Ib ~ Ⅲb with complete resection, chemotherapy is performed in 6 weeks after resection, including tumor size > 2cm of stage Ia;
6. Blood routine: N > 1.5×109/L、PLT > 100×109/L, normal liver function and kidney function;
7. Voluntarily involved to clinical study and sign informed consent.

Exclusion Criteria:

1. Suffering from other primary malignant tumor in 5 years;
2. Incomplete resection or uncertain to take resection;
3. Serious disease of heart, liver, kidney with severe dysfunction;
4. Pregnancy or breast-feeding women;
5. Mental or cognitive disorders which would influence judgment of QOL in this study;
6. During or had adjuvant chemotherapy;
7. Being participating other drug trials;
8. Allergy to the drug in our study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
quality of life（QoL) | every three weeks

SECONDARY OUTCOMES:
two-year disease-free survival rate and disease-free survival | once every three months

CONTACTS AND LOCATIONS:
Overall Officials: xu ling, Principal Investigator — Shanghai University of Traditional Chinese Medicine; xu ling, doctor, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - ShanghaiUTCM, Shanghai, Shanghai Municipality
  - Xuling, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Wang Y, Jiao L, Chen Z, Xu J, Che J, Huang H, Zhang L, Shen X, Yang Y, Zhao T, Zhang J, Zhou D, Wang Q, Yao J, Yang W, Sun C, Li J, Bi L, Ding R, Goodfellow I, Gong Y, Xu L. Adjuvant Chemotherapy with Traditional Chinese Herbal Granules Versus Placebo in Resected Non-Small Cell Lung Cancer: Updated Survival Analysis of a Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Integr Cancer Ther. 2026 Jan-Dec;25:15347354251409081. doi: 10.1177/15347354251409081. Epub 2026 Jan 27. PMID 41589575
- [Derived] Wang Q, Jiao L, Wang S, Chen P, Bi L, Zhou D, Yao J, Li J, Wang L, Chen Z, Jia Y, Zhang Z, Shen W, Zhu W, Xu J, Gao Y, Xu L, Gong Y. Adjuvant Chemotherapy with Chinese Herbal Medicine Formulas Versus Placebo in Patients with Lung Adenocarcinoma after Radical Surgery: a Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. Biol Proced Online. 2020 Mar 1;22:5. doi: 10.1186/s12575-020-00117-5. eCollection 2020. PMID 32140080
- [Derived] Xu L, Li H, Xu Z, Wang Z, Liu L, Tian J, Sun J, Zhou L, Yao Y, Jiao L, Su W, Guo H, Chen P, Liu J. Multi-center randomized double-blind controlled clinical study of chemotherapy combined with or without traditional Chinese medicine on quality of life of postoperative non-small cell lung cancer patients. BMC Complement Altern Med. 2012 Aug 1;12:112. doi: 10.1186/1472-6882-12-112. PMID 22853619